CLINICAL TRIAL: NCT03321227
Title: Effect of Eggs and Egg Components on Cognitive Performance and Appetite in School-aged Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Nick Bellissimo, Associate Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Ryerson-REB-2017
Record Dates: First submitted 2017-10-18; First posted 2017-10-25 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Nutrition; Cognitive Performance; Appetite
Keywords: Children; Nutrition; Eggs; Cognitive performance; Glycemic response; Appetite; Emotion
MeSH Terms: interventions — Egg White; Egg Yolk; Yogurt

STUDY DESIGN:
Intervention Model Description: A random and within subject repeated measures experiment to study the effects of egg consumption on cognitive performance in children and the underlying physiological mechanisms in this relationship.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Snack skipping (Experimental): No snack provided
  Interventions: Other: Snack skipping
- Whole eggs (Experimental): 2 whole large eggs as a snack
  Interventions: Other: Whole eggs
- Egg whites (Experimental): 2 egg whites as a snack
  Interventions: Other: Egg whites
- Egg yolks (Experimental): 2 egg yolks as a snack
  Interventions: Other: Egg yolks
- Yogurt (Active Comparator): Full fat yogurt as a snack
  Interventions: Other: Yogurt

INTERVENTIONS:
Other: Snack skipping — No snack provided
  Arms: Snack skipping
Other: Whole eggs — 2 whole large eggs scrambled, provided as a snack
  Arms: Whole eggs
Other: Egg whites — 2 egg whites scrambled, provided as a snack
  Arms: Egg whites
Other: Egg yolks — 2 egg yolks scrambled, provided as a snack
  Arms: Egg yolks
Other: Yogurt — A serving of full fat yogurt that is isocaloric to the 2 whole eggs
  Arms: Yogurt

SUMMARY:
The purpose of the present study is to determine the effects of eggs and egg components on cognitive performance and appetite in children aged 9-14 years, as well as to identify the underlying physiological mechanisms in this relationship.

DETAILED DESCRIPTION:
Children will be asked to refrain from exercising the morning of their test day and inform researchers of any illness. Following a 12-hour overnight fast, children will consume a standardized breakfast of a cereal bar, fruit cup and orange juice at home (total 330 kcal). Children will be asked to avoid consumption of any other food, with the exception of water, until arrival at the laboratory 3 hours later.

At the laboratory, five treatments of: (a) 2 whole eggs, (b) 2 egg whites, (c) 2 egg yolks, (d) full fat yogurt isocaloric to the 2 whole eggs, and (e) snack skipping will be provided to children 9-14 years on separate days at least 7 days apart. Cognitive performance, subjective emotion/mood, and subjective appetite will be measured for 90-minutes following snack consumption (n=25). Cognitive performance assessments will include learning and memory, spatial memory, attention and processing speed, and executive functions. In a subgroup of individuals (n=10), glucose, insulin, incretin hormones (glucagon like peptide1(GLP1) and gastric inhibitory polypeptide (GIP)),dipeptidyl peptidase 4 (DPP4), amino acids, fatty acids, and choline will be measured for 90-minutes following snack consumption.

ELIGIBILITY:
Inclusion Criteria:

* be between 9 and 14 years of age
* be healthy, and have been born at term
* healthy body weight (between the 5th and 85th BMI percentile for age and gender)

Exclusion Criteria:

* children with food sensitivities or allergies to eggs, egg-products, dairy and wheat
* children with any diagnosed learning, emotional, or behavioral disabilities
* children on medications that may influence cognitive performance

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change in memory from baseline | 15, 30, 60, and 90 minutes
  One of five word lists composed of 15 words will be audio-visually presented to children. The majority of the words will be one syllable, and four words in each list will be two syllables long. The list will be presented at baseline and the children will be asked to recall as many words as possible at each time-point. The list will be presented for 2.5 minutes, and children will have 2 minutes for both immediate and delayed recall.
Change in spatial working memory from baseline | 0, 15, 30, 60, and 90 minutes
  Assessed using a spatial pattern recognition test via the Membrain application. The test consists of a series of subtests where children will be presented a picture with patterns to study, and asked to identify a picture with the same pattern from a group of four images. This test will be at each time-point and takes approximately 1 minute to complete.
Change in attention from baseline | 0, 15, 30, 60, and 90 minutes
  The continuous performance task (CPT) will be completed via the Membrain application. During the CPT task, children will be given a sequence of two letters to identify; for example respond to the detection of the letter "X" only when it is preceded by the letter "A". This task will be at each time-point and will take 3 minutes total to complete.
Change in executive function from baseline | 0, 15, 30, 60, and 90 minutes
  The Stroop task will be completed via the Membrain application. Children will be presented with a list of words presented in colors that match the word (congruent, the word 'red' presented in red) or colors that do not match the word (incongruent, the word 'red' presented in blue). Children will be asked to identify the color of the word, not the word itself. The task is scored for the number of correct and incorrect colors identified, as well as total time to completion. This test will be at each time-point and will take 1 minute to complete.

SECONDARY OUTCOMES:
Change from baseline mood | 0, 15, 30, 60, and 90 minutes
  Measured using visual analogue scale (mm). Each VAS is a 100 mm line where they will place a pencil mark to describe their feelings.These emotions will be seperated into three categories including, subjective emotions (aggressive, angry, excited, disappointed, and frustrated), global vigour and affect (alert, sad, tense, effort, happy, weary, calm and sleepy), and wellness. These sub scales will be combined to compute an average total score for each category.
Change from baseline subjective appetite | 0, 15, 30, 60, and 90 minutes
  Measured using visual analogue scale (mm). Each VAS is a 100 mm line where they will place a pencil mark to describe their feelings. Average appetite will combine four questions (desire to eat, hunger, fullness, and prospective food consumption) to calculate the score.
Change from baseline cholecystokinin (CCK) | 0, 15, 30, 60, and 90 minutes
  Blood CCK (pmol/L). CCK concentration in serum will be determined in duplicate via enzymelinked immunosorbent assay kits (ELISA; Millipore, Billerica, Massachusetts).
Change from baseline dipeptidyl peptidase 4 (DPP4) | 0, 15, 30, 60, and 90 minutes
  Blood DPP4 (ng/mL). DPP4 concentration in serum will be determined in duplicate via enzymelinked immunosorbent assay kits (ELISA; Millipore, Billerica, Massachusetts).
Change from baseline glucagonlike peptide1 (GLP1) | 0, 15, 30, 60, and 90 minutes
  Blood GLP1 (pmol/L). GLP1 concentration in serum will be determined in duplicate via enzymelinked immunosorbent assay kits (ELISA; Millipore, Billerica, Massachusetts).
Change from baseline insulin | 0, 15, 30, 60, and 90 minutes
  Blood insulin (pmol/L). Insulin concentration in serum will be determined in duplicate via enzymelinked immunosorbent assay kits (ELISA; Millipore, Billerica, Massachusetts).
Change from baseline glycemic response | 0, 15, 30, 60, and 90 minutes
  Blood glucose will be measured in whole blood using YSI 2300 STAT PLUS (YSI Incorporated, Yellow Springs, OH)
Change from baseline amino acids | 0, 15, 30, 60, and 90 minutes
  From plasma blood samples. Amino acids will be determined using the pre-column derivatization HPLC procedure. A plasma sample will be de-proteinizied with a 5-sulfosalicyclic acid solution, then centrifuged at 4°C and 18,400 G for 15 minutes. The amino acids will be derivatized from the sample with ortho-phthaldehyde reagent. The sample will then be analyzed using the Perkin Elmer Series HPLC System in the Ryerson University Analytical Centre.
Change from baseline fatty acids | 0, 15, 30, 60, and 90 minutes
  From plasma blood samples. Fatty acids will be assessed via gas chromatography, an effective method to measure both the proportions and concentrations of fatty acids in plasma. A plasma sample will be prepared by trans-esterification of total lipid aliquots with a MeOH/HCl mixture and n-hexane. The sample will then be analyzed using the Perkin Elmer Auto-System in the Ryerson University Analytical Centre.
Change from baseline choline | 0, 15, 30, 60, and 90 minutes
  From plasma blood samples. Will be analyzed for choline using a fluorimetric assay; free choline will be oxidized by choline oxidase to betaine and H2O2 that reacts with a specific dye to form a pink colored product. The fluorescence intensity at 530/585 nm is directly proportional to the choline concentration in the sample.

CONTACTS AND LOCATIONS:
Overall Officials: Nick Bellissimo, PhD, Principal Investigator — Toronto Metropolitan University
Locations (1):
- School of Nutrition, Ryerson University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided